CLINICAL TRIAL: NCT01782456
Title: Tolerance of an Oral Nutritional Supplement(ONS)With a New Protein Blend in Healthy Children
Brief Title: Tolerance of an Oral Nutritional Supplement(ONS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AL09
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Gastro-Intestinal Tolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Oral Nutritional Supplement (Experimental): 2 servings per day of a complete and balanced, ready-to-drink oral nutritional supplement with a new protein blend.
  Interventions: Other: Study Oral Nutritional Supplement

INTERVENTIONS:
Other: Study Oral Nutritional Supplement — Supplement contains a new protein mix consisting of a blend of milk, soy, and pea protein.

SUMMARY:
The objective of this study is to capture information on gastrointestinal tolerance (GI) of an oral nutritional supplement containing a new protein blend in healthy children aged ≥ 3 to ≤ 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 3 and ≤ 10 years of age
* Healthy and not suffering from any physical disability.
* Height-for-age and BMI-for-age between the 5th and the 95th percentile as well as a weight-for-age between the 5th and the 85th percentile
* Consumption of 2 servings/day of the investigational product for 7 consecutive days
* Willingness to follow the study procedures and record the data in the diary and complete any forms or assessment as needed throughout the study
* Agreement to not consume a nutritional product that is not study product during the study period

Exclusion Criteria:

* History of an acute or chronic condition that may affect feeding habits or nutritional status
* Medications or nutritional supplements, taken on a daily basis for more than 2 weeks during the past month prior to screening visit that may profoundly affect feeding habits or nutritional status
* Clinically significant nutritional deficiency requiring specific treatment
* Acute/chronic condition requiring medical treatment which may include hospitalization such as diabetes or stress induced hyperglycemia, dialysis treatment, inflammatory bowel disease, pancreatitis, autoimmune disease or immunodeficiency, celiac disease, cystic fibrosis, active tuberculosis, malformation of the gastrointestinal tract or gastroesophageal reflux disease
* History of constipation
* Allergy or intolerance to any ingredient in the study product
* Gastrointestinal infection or acute diarrhea at the time of study start
* Hepatitis B or C, or HIV, or malignancy
* Congenital cardiac defects
* Antibiotic therapy within last 2 weeks of start of study
* Dysphagia, aspiration risk, difficulty in swallowing due to acquired/congenital abnormalities

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2013-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Gastro-Intestinal Tolerance | Study Day 1-7
  Self-reported Questionnaire

SECONDARY OUTCOMES:
Study Supplement Compliance | Study Day 1-7
  Self-reported number of servings consumed per day
Weight | Study Day 1 and 8
Height | Study Day 1 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Williams, MPH, Study Chair — Abbott Nutrition
Locations (1):
- Radiant Research, Inc., Cincinnati, Ohio, United States